CLINICAL TRIAL: NCT05537077
Title: Comparison of Effectiveness of Dextrose Prolotherapy Treatment With Different Concentrations in Patients With Knee Osteoarthritis
Brief Title: Different Concentrations of Dextrose Prolotherapy Treatment in Knee Osteoartritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turkish League Against Rheumatism (Other)
Responsible Party: Principal Investigator, Muhammet Uğur ÖZTÜRK, Medical Doctor, Turkish League Against Rheumatism
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRASD-MUO-TEZ
Record Dates: First submitted 2022-09-03; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Prolotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): %5 Dextrose prolotherapy, hotpack therapy and home based exercise program was applied to group 1.
  Interventions: Other: Prolotherapy; Other: Home based exercise program; Other: Hotpack therapy
- Group 2 (Active Comparator): %10 Dextrose prolotherapy, hotpack therapy and home based exercise program was applied to group 2.
  Interventions: Other: Prolotherapy; Other: Home based exercise program; Other: Hotpack therapy
- Group 3 (Active Comparator): %20 Dextrose prolotherapy, hotpack therapy and home based exercise program was applied to group 3.
  Interventions: Other: Prolotherapy; Other: Home based exercise program; Other: Hotpack therapy
- Group 4 (Active Comparator): Hotpack therapy and home based exercise program was applied to group 4.
  Interventions: Other: Home based exercise program; Other: Hotpack therapy

INTERVENTIONS:
Other: Prolotherapy — DPT was applied as a total of 3 sessions at 0, 3 and 6 weeks. In each session, intra-articular 5 ml and periarticular 10 ml dextrose injections were administered to the knee. Periarticular injection was applied to 10 points as 1 ml in each region. The regions were determined as medial and lateral coronary ligaments, proximal and distal medial and lateral collateral ligaments, pes anserinus region, proximal and distal patellar tendon, quadriceps tendon attachment area.
  Arms: Group 1; Group 2; Group 3
Other: Home based exercise program — Knee ROM, isometric and isotonic quadriceps strengthening exercises were given as 2 sets of 10 repetitions per day for 12 weeks.
Other: Hotpack therapy — Hotpack treatment was applied for 20 minutes at 0, 3 and 6 weeks.

SUMMARY:
In this study, the investigators aimed to compare the efficacy of %5, %10 and %20 concentration dextrose prolotherapy (DPT) treatments in patients with primary knee osteoarthritis (OA). In this prospective, randomized, controlled, single-blind study, 128 patients who met the inclusion criteria were recruited and divided into four groups. Thirty patients from each group completed the study. %5 DPT was applied to Group 1, %10 to Group 2, and %20 to Group 3 in combination with home exercise program and hotpack therapy. Group 4 was given home exercise program and hotpack therapy. Groups were evaluated with VAS (Visual Analog Scale), WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index), knee ROM (Range of Motion), and Timed up and go test (TUG) parameters. DPT groups were evaluated in terms of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-70 years,
* Knee pain for more than three months,
* Diagnosed with primary knee OA according to ACR clinical/radiological diagnostic criteria and Kellgren-Lawrence stage II-III.

Exclusion Criteria:

* Total knee replacement
* Rheumatological diseases, systemic infection, and malignancy
* Pregnancy or breastfeeding
* Taking a nonsteroidal anti-inflammatory drug (NSAID) in the last week, taking steroid drugs in the last month
* Undergoing anticoagulant or immunosuppressive therapy
* Knee injection in the last 6 months

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) | Pre-intervention, sixth week, twelfth week.
  VAS is a scale used to evaluate pain severity. Pain severity is evaluated between 0 and 10. A high score indicates a bad result.
Change in Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC) | Pre-intervention, sixth week, twelfth week.
  WOMAC; It consists of three subcategories: pain, stiffness, and physical function difficulty. A score of 20 for pain, 8 for stiffness, 68 for physical function difficulty, and a total of 96 points can be obtained. An increase in the score is interpreted as more pain, stiffness and loss of function.
Change in Knee Joint Range of Motion | Pre-intervention, sixth week, twelfth week.
  Knee flexion in the prone position and knee extension in the supine position were measured actively and passively with a goniometer.
Change in The Timed "Up & Go" Test | Pre-intervention, sixth week, twelfth week.
  In this test, balance, walking speed and functional capacity are evaluated. Patients who complete the test in less than 10 seconds are considered independent.

SECONDARY OUTCOMES:
Change in Short Form 36 (SF-36) | Pre-intervention, twelfth week.
  SF-36 used for determining quality of life. It consists of eight sub-parameters such as physical functioning, role physical, mental health, role emotional, bodily pain, social functioning, vitality and general health and a total of 36 questions. Each parameter is scored between 0 and 100. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Faculty of Medicine, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wee TC, Neo EJR, Tan YL. Dextrose prolotherapy in knee osteoarthritis: A systematic review and meta-analysis. J Clin Orthop Trauma. 2021 May 20;19:108-117. doi: 10.1016/j.jcot.2021.05.015. eCollection 2021 Aug. PMID 34046305
- [Background] Sert AT, Sen EI, Esmaeilzadeh S, Ozcan E. The Effects of Dextrose Prolotherapy in Symptomatic Knee Osteoarthritis: A Randomized Controlled Study. J Altern Complement Med. 2020 May;26(5):409-417. doi: 10.1089/acm.2019.0335. Epub 2020 Mar 30. PMID 32223554
- [Derived] Ozturk MU, Baygutalp F. A comparative analysis of prolotherapy efficacy in patients with knee osteoarthritis across varied dextrose concentrations. Clin Rheumatol. 2023 Dec;42(12):3321-3331. doi: 10.1007/s10067-023-06723-4. Epub 2023 Aug 4. PMID 37540383